CLINICAL TRIAL: NCT04978844
Title: The Bio-psycho-social Effects of a Novel Form of Psychotherapy for Preschool Children Suffering From Anxiety Disorders: a Comparison of Short-term Play Therapy, Dyadic Therapy and Controls
Brief Title: A Brief Emotion Focused Therapy for Preschoolers With Anxiety Disorders
Acronym: I-WotCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Interdisciplinary Center Herzliya (Other)
Responsible Party: Principal Investigator, Yael Apter, Research psychologist, Interdisciplinary Center Herzliya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Inner World of the Child
Record Dates: First submitted 2021-07-17; First posted 2021-07-27 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Childhood Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: I-WotCH, Dyadic and Controls
Who Masked: Outcomes Assessor
Masking Description: outcome assessors: Post graduate students in clinical psychology, lab technicians
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- I-WotCH (Active Comparator): I-WotCH- Inner World of the Child- is a novel innovative therapy developed in our clinic. The therapy is based on modern concepts of early childhood developments emphasizing themes related to emotional regulation, processes of socialization, observational research on interpersonal and behavior as well as recent developments on affiliative neuroscience. More specifically, the therapist, through play, identifies themes and emotions the child is preoccupied with. The therapist then assists the child in naming these emotions, validating them, exploring their nature and consequences. The therapists discussed ways of managing and self-regulating these emotions. These methods would include behavioral techniques, the ability to enlist help from others and reframing. In addition, the therapy will address dealing with complexed emotions and enhancing symbolic play and joyfulness.
  Interventions: Behavioral: IWOTCH
- Dyadic therapy (Active Comparator): Child parent psychotherapy: CPP consists of joint parent-child sessions that focus on the child's free play and spontaneous parent-child interaction. The CPP therapist acts to "translate" the developmental and emotional meaning of a child's emotions and actions to the parent. The target of treatment includes the both the child's and the caregiver's adaptive conflicts, including a parent's difficulty in providing sensitive and developmentally appropriate care. CPP fosters parent-child activities that foster mutual pleasure, interpersonal trust and understanding. In the purpose of this study only mothers will be included.
  Interventions: Behavioral: Dyadic therapy
- Control (No Intervention): Healthy control.

INTERVENTIONS:
Behavioral: IWOTCH — Arm 1
  Arms: I-WotCH
Behavioral: Dyadic therapy — Arm 2
  Arms: Dyadic therapy

SUMMARY:
The study will comprise of three groups of children (n=40): 1. A group receiving a novel short-term dynamic play therapy. 2. Dyadic therapy 3. Control group who will not receive therapy. All children will be assessed for psychopathology (anxiety, depression and behavioral problems) using standardized instruments such as semi-structured interview and self-reported questionnaires; EEG recordings will be performed from child and parents in order to asses brain synchrony; Cortisol (CT), Dehydroepiandrosterone (DHEA), Oxytocin (OT) and Secretory Immunoglobulin A (SIgA) will be assessed by using saliva sampling; and father-mother-child interactions will be videotaped and analyzed. Narrative descriptions will be obtained from parents, and the interviews recorded for voice analysis. Assessment will be made at baseline and then bi-monthly for six months.

DETAILED DESCRIPTION:
Anxiety disorders are the most common disorders across the lifespan and tend to have both an early onset and persistent course throughout life. Since the preschool years mark a sensitive period for the development and exacerbation of anxiety symptoms in children, which often persist throughout childhood and adolescence, there is an urgent need to understand this condition in the most detailed manner and find efficient therapeutic solutions. In this Randomized control study (RCT), the investigators will test the efficacy of two interventions for childhood anxiety disorders: a special emotion-focused therapy and a dyadic parent-child intervention.

DESGIN Recruitment: consecutive admissions to the preschool clinic at the Intradisciplinary Center at Herzliya will be asked to participate in the study.

Baseline Diagnosis:

1. Psychiatric diagnosis: will be made by using a combination and integration of the childhood version of the Schedule for Schizophrenia and Affective Disorders (K-SADS-PL) and the Preschool Age Psychiatric Assessment (PAPA). Diagnosis will be made according to the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) and Diagnostic Classification of Mental Health and Developmental Disorders of Infancy and Early Childhood (DC 0-5). These semi-structured interviews will be conducted by a clinical psychologist with a special expertise in evaluation and treatment in preschool children (YAL). All diagnoses will then be checked with a senior child and adolescent psychiatrist.
2. Behavioral profiles: The Child Behavioral Checklist for preschoolers will be administered to parents and will generate behavioral profiles adjusted for gender.

Randomization:

Consecutive referrals to the clinic will be recruited for the study and will be randomly and blindly allotted to each treatment arm.

Therapy:

Both therapies would have the same duration of 6 months and will consist of 24 weekly meetings for the child or child-parent dyad, accompanied by 12 bi-weekly meetings with both parents. Each session will last for approximately 50 min.

1. Inner World of the Child I-WotCH- - is a novel innovative therapy developed in our clinic. The therapy is based on modern concepts of early childhood developments emphasizing themes related to emotional regulation, processes of socialization, observational research on interpersonal and behavior as well as recent developments on affiliative neuroscience. More specifically, the therapist, through play, identifies themes and emotions the child is preoccupied with. The therapist then assists the child in naming these emotions, validating them, exploring their nature and consequences. The therapist discusses ways of managing and self-regulating these emotions through methods that include behavioral techniques, the ability to enlist help from others, and reframing. In addition, the therapy will address ways of dealing with complex emotions and enhancing symbolic play and joyfulness
2. Child-parent psychotherapy- CPP: CPP consists of joint parent-child sessions that focus on the child's free play and spontaneous parent-child interaction. The CPP therapist acts to "translate" the developmental and emotional meaning of a child's emotions and actions to the parent. The target of treatment includes the both the child's and the caregiver's adaptive conflicts, including a parent's difficulty in providing sensitive and developmentally appropriate care. CPP fosters parent-child activities that foster mutual pleasure, interpersonal trust and understanding. In the purpose of this study only mothers will be included.

EVALUATION All children will be evaluated at baseline, at bi-monthly intervals during treatment, and at termination (at 6 months). The evaluation session will be conducted in a university laboratory (not in the clinical setting) by RA unfamiliar to the child.

Dropouts will be noted and as far as possible the details for discontinuing will be recoded.

1. Psychopathology (as noted above):

1. Psychiatric diagnosis: will be made by using a combination and integration of the K-SADS-PL and the PAPA. Diagnosis will be made according to the DSM-5 and DC 0-5.
2. Behavioral profiles: The Child Behavioral Checklist for preschoolers will be administered to parents.

2. Parent-Child Relationship:

1. Parent-Child Social Interactions: each five minutes of mother-child, father-child and triadic interactions with pre-selected toys will be videotaped. Dyadic interaction will include free play and a challenging task. Interactions will be coded with the Coding Interactive Behavior manual. The CIB is a global rating system for analyzing social interactions between two or more partners. The CIB comprises five manuals: newborns, infants, preschoolers, adolescents/ adults, and the recently added psychotherapy manual, all based on the same constructs with good psychometric properties. The CIB utilizes a variety of social settings and observational paradigms (e.g., free play, feeding, conflict discussion, triadic/family interactions) and has been used in hundreds of published studies in healthy and high-risk populations and clinical trials.

   The following dimensions will be emphasized:
   1. Iintrusiveness- this measures the degree to which the parent interferes with the child's natural behavior throughout the session, for instance, ignoring the child's signals, overriding the child's cues and wishes.
   2. Reciprocity: this measures the degree to which the parent and child interact in a mutual fashion.
   3. Acknowledgment: this scale is a central feature of sensitive parenting. this measures the degree to which the parent is aware and sensitive to child's signals and expresses them both vocally and by gesture.
   4. Avoidance- this measures the degree to which the child avoids the parent and retreats from the parent's attempts to engage him.
   5. Positive and negative affect: this measures the degree to which the parent expresses positive or negative emotions towards the child.

   In addition, other dimensions will also be noted and scored, as listed in the CIB manual.
2. Mother-Father Relationship: five minutes of Conflictual Discussion between and father will be videotaped and coded.

   3. Child Emotion Regulation: the child's ability to regulate his emotions will be rated using the child's reaction to a challenging task, such as the puzzle task. Micro-coding of child behavior during the puzzle task paradigm will be conducted on a computerized system (Noldus Co, Waggeniggen, The Netherlands). Codes are based on our own and others' research with preschoolers . Child's Self-Regulation will be represented by the sum of time proportions of each of the following behaviors: withdrawal, gaze aversion, physical self-soothing and solitary substitutive play.

   In addition, parents will fill out the Toddler Behavior Assessment Questionnaire (TBAQ), . This questionnaire includes the assessment of child's temperament, emotion regulation, self-soothing and inhibition control.

   4. Parental Representation of Child and the Treatment: Narrative descriptions will be obtained from parents, and the interviews recorded for voice analysis. Parents will answer three questions: 1. "Describe your child"; 2. "Describe your child's problems"; 3. "How do you think the therapy will help addressing your child's difficulties".

   5. Biological Measures:

   1. Hormonal Measures: Saliva will be obtained for the following measure for both parents and child: OT, CT and DHEA (DHEA from parents only).

   OT: Oxytocin is a hormone which appears to be a marker of affiliation and relationship. It has been shown to be disturbed in conditions where parent-child relationships are impaired.

   CT: is a well known and much studied marker of stress and anxiety. DHEA: this hormone has also been shown by our group and others to be related to stress and emotional regulation.

   Hormonal Analysis:

   OT: The liquid samples will be stored at 80ºC. To concentrate samples by 3 or 4 times, the liquid samples would be lyophilized over-night and kept in 20ºC until assayed. Dry samples will be reconstructed in the assay buffer immediately before analysis by EIA. Determination of OT was performed by commercial OT ELISA kit (Assay Design, MI, USA).

   CT: The samples will be stored at -20°C until assayed. Cortisol levels will be assayed using a commercial ELISA kit (Assay Design, MI).

   DHEA: In-order to precipitate the saliva, samples will undergo several freeze-thaw cycles. After the fourth cycle the tubes will be centrifuged at 1500 x g (@3000 rpm) for 20 minutes. Supernatants will be stored at -20°C until assayed. Determination of DHEA will be performed using a commercial DHEA ELISA kit (Salimetrics, USA). Salimetrics DHEA kit is a competitive immunoassay specifically designed for the quantitative measurement of salivary DHEA. On the day of assay, samples will be thawed, and 50 micro-liters will pipette into the appropriate well of the kit.

   Immunological measures:

   SIgA: there is a strong relationship between the immunological system and stress. the investigators will therefore assay SIgA, which has also been studied in stressful situations.

   Immunological measure analysis:

   Determination of s-IgA will be performed using a commercial s-IgA ELISA kit (EUROIMMUN AG: 23560, Luebeck, Germany). The kit provides quantitative in vitro assay for s-IgA in human saliva. On day of assay, samples will be thawed completely and diluted 1:201 in sample buffer and further measured according the kit's instructions. Measurements were performed in duplicate and the concentrations of samples were calculated by using matrix laboratory (MATLAB 7) according to relevant standard curves. The intra-assay coefficient of samples and controls was 8.1%, and inter-assay coefficients for samples and controls were less than 11.6%.

   Electrophysiological measure:

   EEG recordings will be performed on the first and final visit. Children and parents will be given an EEG helmet from which multiple scalp readings will be taken.

   Statistics all variables will be entered into a data base and then into SPSS. The major hypothesis will be the relative efficacy of the two interventions would be compared to control, evaluating symptoms reduction, hormonal level changes and enhancing parental sensitivity (among other changes in parental behavior). The investigators will perform variance analysis, correlations, regression and HLM models that will describe the changes in these variables in each group (two intervention and one control) along the check up points (baseline, every two months and at ending point).

ELIGIBILITY:
Inclusion Criteria:

All consecutive admission to the early childhood clinic at the IDC Herzliya

Exclusion Criteria:

Parents and children not living in the same household

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Symptom change as measured by the CBCL | Every two months for a period of six months
  The CBCL measures symptoms of psychopathology in a quantitive manner. Reduction in the number symptoms means a favorable outcome.
Maternal Sensitivity as measured with the CIB (coding interactional behavior) | Every two months for a period of six months
  This measure is a video of mother-child interactions, a higher score is a more favorable outcome. scores range from a minimum of 0 to a maximum of 5.

CONTACTS AND LOCATIONS:
Overall Officials: Feldman Ruth, Prof, Principal Investigator — IDC Herzliya
Locations (1):
- The Preschool clinic at the Interdisciplinary Center Herzlyia, Herzliya, Select A State Or Province, Israel